CLINICAL TRIAL: NCT03994133
Title: Contribution of Body Composition Monitor (BCM) Among Patients Using Daily Home Dialysis With Low Dialysate Flow : French Study Cohort
Brief Title: Body Composition Monitor Among Daily Home Dialysis With Low Flow Dialysate
Acronym: VOLODIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03451-54
Record Dates: First submitted 2019-06-14; First posted 2019-06-21 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-07

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Hemodialysis, Home; Electric Impedance
Keywords: Dialysis; BCM; Daily Home Dialysis; low-flow dialysate; Fluid Overload; kt/V; dialysis dose; Nutritional Status; blood pressure
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Daily Home Dialysis patients: Daily Home Dialysis patients with low-flow dialisate for more than 3 months in France
  Interventions: Other: Measurement of the hydration state by bio-impedance spectroscopy

INTERVENTIONS:
Other: Measurement of the hydration state by bio-impedance spectroscopy — * The measurements will be performed in each center by a reference physician or nurse, using a portable whole body bioimpedance spectroscopy device, BCM (Fresenius Medical Care).
  * The electrodes will be attached to one hand and one foot on the ipsilateral side, after the patient has been in the supine position for at least 5 minutes.
  * The measurement will be done in pre-dialytic

SUMMARY:
The fluid overload measured by the Body Composition Monitor (BCM Fresenius Medical Care) is a new independent risk factor of mortality.

This risk has already been described in intermittent hemodialysis patients and peritoneal dialysis patients but never evaluated in Daily Home Dialysis with low dialysate flow.

The investigator propose a first study measuring the state of hydration by impedancemetry (BCM) in this population.

The aim of this work is to to analyze hydration status in a representative sample of prevalent Daily Home Dialysis with low-flow Dialysate patients.

Secondary objectives are to identify associations between hydration status and patient characteristics and treatment practice in order to find out which conditions should alert the clinician to potential fluid overload, to compare these results with the peritoneal dialysis population and in center hemodialysis population, to evaluate the correlation between impedancemetry and blood pressure in this population, to assess the nutritional status and evaluation of a new method of measurement of kt / V based on impedancemetry, without recourse to a blood test.

DETAILED DESCRIPTION:
Study objectives

This study is a cross sectional, observational trial in 11 centers in France. The primary objective is to analyze hydration status in a representative sample of prevalent Daily Home Dialysis with low-flow Dialysate patients.

Secondary objectives are to identify associations between hydration status and patient characteristics and treatment practice in order to find out which conditions should alert the clinician to potential fluid overload, to compare these results with the peritoneal dialysis population and in center hemodialysis population, to evaluate the correlation between impedancemetry and blood pressure in this population, to assess the nutritional status and evaluation of a new method of measurement of kt / V based on impedancemetry, without recourse to a blood test.

Centers

Participants in this study are: CHU de Caen, Tenon Hospital, CHG Saint-Lô, CHG Alençon, CHG Flers, CHG Lisieux, CHG Evreux, ANIDER Rouen, CHG Le Havre, A.U.B Rennes, A.D.P.C Marseille.

Patients

In each center, all prevalent patients, for more than 3 months, on Daily Home Dialysis with Low-flow Dialysate are assessed for eligibility for inclusion if they are older than 18 years of age and want to sign informed consent. Patients are excluded if they have a cardiac pacemaker or metallic implants, are amputees or are pregnant. Patients are evaluated during a routine clinical visit. All patients will signed informed consent, and ethical advice is obtained.

Measurements of hydration and body composition

BCM measurements will be performed in each center by one reference physician or nurse, using a portable whole body bioimpedance spectroscopy device, the BCM (Fresenius Medical Care). The BCM measures the impedance spectroscopy at 50 different frequencies between 5 kHz and 1 MHz. The BCM was validated intensively against all available gold-standard methods.

The measurement will be performed in pre-dialysis, electrodes will be attached to one hand and one foot at the ipsilateral side, after the patient will be in recumbent position for at least 5 minutes. Reproducibility of BCM derived parameters is high, with a coefficient of variation for the interobserver variability ECW and TBW around 1.2%. Therefore, only one BCM measurement is performed in each individual patient.

Extracellular water (ECW), intracellular water (ICW) and total body water (TBW) are determined from the measured impedance data following the model of Moissl et al en 2006.

Fluid overload is expressed by a compartment called OH (overhydration). OH represents the difference between the amount of ECW in the tissue as actually detected by the BCM and the amount of water present in tissue, as predicted by physiological models under normal physiological (normohydrated) conditions. Of note, OH has no direct relation to circulating volume.

Four hydrations groups are defined, based on studies by Wieskotten et al. on healthy population and Wabel et al. on a dialysis population: Normohydrate group: OH between -1.1L and + 1.1L (corresponding to the 10th and 90th percentiles of a population of the same gender distribution and with a comparable age band out of a healthy reference cohort, where hydration status was measured with the identical technology); Hypovolemic group: OH <-1.1L; Fluid overload group: OH between + 1.1L and + 2.5L; Severe fluid overload group: OH> + 2.5L.

The post-dialysis OH status will be obtained by the difference between pre-dialysis OH obtained by impedancemetry and the UF performed.

Blood pressure will be performed in pre-dialytic and post-dialytic and is recorded as the mean of two consecutive measurements with 5 minutes interval, using one single calibrated device in each center. The investigator defined 3 groups according to pre-dialysis systolic blood pressure (SBP): Hypertensive: SBP > 140 mmHg; Normotendu: SBP [100-140 mmHg]; Hypotensive: SBP < 100 mmHg.

Height and weight will be measured using one single calibrated device in each center.

Clinically relevant parameters will be registered in the case report form (CRF).

Nutritional assessment

Nutritional status is evaluated using three methods:

The first one is The Mini Nutritional Assessment (MNA), on 30 points, is a questionnaire of 18 questions to define three groups: 24-30 points: normal nutritional status; 17-23.5 points: risk of malnutrition and < 17 points: poor nutritional status.

The second one is the Scale of Assessment of the food intake (EPA) is a rapid tool based on self-assessment by analog scale from 0 to 10. An EPA> 7 should result in nutritional management.

The third is according to the impedancemetry. The BCM (Fresenius Medical Care), provides, according to Chamney et al. Model, two parameters: "LTM" and "FTM" for "lean tissue mass" and "fat tissue mass". The values obtained will be normalized to the body surface, to allow a comparison between patients of different size, thus giving the lean tissue index (LTI = LTM / height2) and the fat tissue index (FTI = FTM / height2). The values for LTI and FTI will be compared to a healthy reference population matched by age and sex. Values below the 10th percentile of the reference population will be considered clinically significant.

Résults were registered in the case report form (CRF).

Patient characteristics

All this information will be collected using two questionnaires given to one reference physician or nurse and the patient respectively.

The investigator identified diabetes (assumed to be present in patients using glucose lowering drugs or insulin), nephropathy, residual diuresis, comorbidities allowing the calculation of the Charlson score, numbers of antihypertensive drugs, hospitalization less than three months old, history of peritoneal dialysis and / or transplantation.

Concerning the daily practice of home dialysis the investigator identified ultrafiltration, blood flow, length of sessions, type of vascular access and creation date, the usual time of the session, the person performing the fistula puncture at home, needle type, frequent problem with connection, observance of dialysis sessions, date of installation at home The following biochemical parameters will be determined in the local laboratories from blood collected during the routine visit. Predialytic dosage: hemoglobin, hematocrit, platelets, leukocytes, urea, creatinine, serum iron, CST, ferritin, sodium, chlorine, potassium, magnesium, alkaline reserve, protidemia, albumin, prealbumin, CRP, PTH, calcium, phosphorus, BNP, B2-microglobulin. Postdialytic dosage: sodium, chlorine, potassium, alkaline reserve, urea, protidemia, B2-microglobulin.

New Kt/V measurement method

Conventionally in dialysis patients, the dialysis dose is represented by the formula kt / V, with: k= plasma clearance of urea; t= unit of time; V= volume of distribution of urea in dialysis patient.

The current assessment is Daugirdas2: Kt / V = -ln (R- (0.008 * t) + ((4 (3.5 * R)) * UF%), with: R= Urea after / Urea before; t= time of the session (hour); UF%= 100*/post-dialysis weight, Our current method therefore requires a plasma dosage of urea at the beginning and end of the session.

The investigator propose a new measurement method where the V will be obtained by impedancemetry and the t corresponds to the duration of the session. For k, the investigator rely on the fact that in vitro (27), at low dialysate flow rate, the saturation of the dialysate in urea is constant, and therefore that the k can be represented by the formula: k = ax Qd (with a: saturation constant and Qd: dialysate flow) Therefore, the investigator propose the following formula: Dialysis dose = a x Qd x t / V This is a new measurement method with important clinical relevance since it avoids two blood tests and two biological tests.

The investigator would therefore like to assume that the measure of kt / V would be equivalent between the formula the investigator would like to test and the conventional formula, either: a x Qd x t / V ≡ kt / V Daugirdas2

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic end stage renal failure
* Patient prevalent in home daily hemodialysis with low dialysate rate for more than 3 months.
* Patient followed at the University Hospital of Caen, Tenon Hospital (Paris), CHG Saint-Lô, CHG Alençon, CHG Flers, CHG Lisieux, CHG Evreux, ANIDER Rouen, CH Le Havre, A.U.B Rennes, A.D.P.C. Marseille

Exclusion Criteria:

* Reversindication to impedancemetry: patient with a pacemaker or an implantable defibrillator,
* Population not validated for impedancemetry: pregnant or lactating woman, major amputation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic end-stage renal disease in home daily hemodialysis with dialysate low for more than three months in France
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
OH sector measurement by bio-impedancemetry. | 5 minutes
  Two electrodes will be glued to one wrist and two others to the ipsilateral ankle. The measurement is painless.
  Distribution of patients in 4 groups:
  Normohydrate group: OH between -1.1L and + 1.1L Hypovolemic group: OH <-1.1L Hyperhydrate group: OH between + 1.1L and + 2.5L Heavy hyperhydrate group: OH> + 2.5L

SECONDARY OUTCOMES:
Measuring blood pressure | 10 minutes
  After 5 minutes of rest, two consecutive measurements at 5 intervals
EPA scale | 1 minutes
  EPA scale is a analogical visual scale of nutrition. Graduated from 0 to 10. 0 = need for nutritional intervention, 10 = good nutritional status
Mini Nutritional Assessment (MNA) score | 5 minutes
  30 points, spread over 18 questions from 24 to 30 points: normal nutritional status from 17 to 23.5 points: risk of malnutrition less than 17 points: poor nutritional status

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] FHN Trial Group; Chertow GM, Levin NW, Beck GJ, Depner TA, Eggers PW, Gassman JJ, Gorodetskaya I, Greene T, James S, Larive B, Lindsay RM, Mehta RL, Miller B, Ornt DB, Rajagopalan S, Rastogi A, Rocco MV, Schiller B, Sergeyeva O, Schulman G, Ting GO, Unruh ML, Star RA, Kliger AS. In-center hemodialysis six times per week versus three times per week. N Engl J Med. 2010 Dec 9;363(24):2287-300. doi: 10.1056/NEJMoa1001593. Epub 2010 Nov 20. PMID 21091062
- [Background] Chertow GM, Levin NW, Beck GJ, Daugirdas JT, Eggers PW, Kliger AS, Larive B, Rocco MV, Greene T; Frequent Hemodialysis Network (FHN) Trials Group. Long-Term Effects of Frequent In-Center Hemodialysis. J Am Soc Nephrol. 2016 Jun;27(6):1830-6. doi: 10.1681/ASN.2015040426. Epub 2015 Oct 14. PMID 26467779
- [Background] Mathew A, McLeggon JA, Mehta N, Leung S, Barta V, McGinn T, Nesrallah G. Mortality and Hospitalizations in Intensive Dialysis: A Systematic Review and Meta-Analysis. Can J Kidney Health Dis. 2018 Jan 10;5:2054358117749531. doi: 10.1177/2054358117749531. eCollection 2018. PMID 29348924
- [Background] Kjellstrand CM, Buoncristiani U, Ting G, Traeger J, Piccoli GB, Sibai-Galland R, Young BA, Blagg CR. Short daily haemodialysis: survival in 415 patients treated for 1006 patient-years. Nephrol Dial Transplant. 2008 Oct;23(10):3283-9. doi: 10.1093/ndt/gfn210. Epub 2008 May 5. PMID 18458034
- [Background] Weinhandl ED, Liu J, Gilbertson DT, Arneson TJ, Collins AJ. Survival in daily home hemodialysis and matched thrice-weekly in-center hemodialysis patients. J Am Soc Nephrol. 2012 May;23(5):895-904. doi: 10.1681/ASN.2011080761. Epub 2012 Feb 23. PMID 22362906
- [Background] Raimann JG, Chan CT, Daugirdas JT, Depner T, Gotch FA, Greene T, Kaysen GA, Kliger AS, Kotanko P, Larive B, Lindsay R, Rocco MV, Chertow GM, Levin NW; Frequent Hemodialysis Network (FHN) Trial Group. The Effect of Increased Frequency of Hemodialysis on Volume-Related Outcomes: A Secondary Analysis of the Frequent Hemodialysis Network Trials. Blood Purif. 2016;41(4):277-86. doi: 10.1159/000441966. Epub 2016 Jan 21. PMID 26795100
- [Background] Kaysen GA, Greene T, Larive B, Mehta RL, Lindsay RM, Depner TA, Hall YN, Daugirdas JT, Chertow GM; FHN Trial Group. The effect of frequent hemodialysis on nutrition and body composition: frequent Hemodialysis Network Trial. Kidney Int. 2012 Jul;82(1):90-9. doi: 10.1038/ki.2012.75. Epub 2012 Mar 28. PMID 22456602
- [Background] Ipema KJ, Struijk S, van der Velden A, Westerhuis R, van der Schans CP, Gaillard CA, Krijnen WP, Franssen CF. Nutritional Status in Nocturnal Hemodialysis Patients - A Systematic Review with Meta-Analysis. PLoS One. 2016 Jun 20;11(6):e0157621. doi: 10.1371/journal.pone.0157621. eCollection 2016. PMID 27322616
- [Background] Weinhandl ED, Nieman KM, Gilbertson DT, Collins AJ. Hospitalization in daily home hemodialysis and matched thrice-weekly in-center hemodialysis patients. Am J Kidney Dis. 2015 Jan;65(1):98-108. doi: 10.1053/j.ajkd.2014.06.015. Epub 2014 Jul 29. PMID 25085647
- [Background] Suri RS, Li L, Nesrallah GE. The risk of hospitalization and modality failure with home dialysis. Kidney Int. 2015 Aug;88(2):360-8. doi: 10.1038/ki.2015.68. Epub 2015 Mar 18. PMID 25786099
- [Background] Finkelstein FO, Schiller B, Daoui R, Gehr TW, Kraus MA, Lea J, Lee Y, Miller BW, Sinsakul M, Jaber BL. At-home short daily hemodialysis improves the long-term health-related quality of life. Kidney Int. 2012 Sep;82(5):561-9. doi: 10.1038/ki.2012.168. Epub 2012 May 23. PMID 22622497
- [Background] Jaber BL, Schiller B, Burkart JM, Daoui R, Kraus MA, Lee Y, Miller BW, Teitelbaum I, Williams AW, Finkelstein FO; FREEDOM Study Group. Impact of short daily hemodialysis on restless legs symptoms and sleep disturbances. Clin J Am Soc Nephrol. 2011 May;6(5):1049-56. doi: 10.2215/CJN.10451110. Epub 2011 Mar 17. PMID 21415315
- [Background] Jaber BL, Lee Y, Collins AJ, Hull AR, Kraus MA, McCarthy J, Miller BW, Spry L, Finkelstein FO; FREEDOM Study Group. Effect of daily hemodialysis on depressive symptoms and postdialysis recovery time: interim report from the FREEDOM (Following Rehabilitation, Economics and Everyday-Dialysis Outcome Measurements) Study. Am J Kidney Dis. 2010 Sep;56(3):531-9. doi: 10.1053/j.ajkd.2010.04.019. Epub 2010 Jul 29. PMID 20673601
- [Background] Cornelis T, Usvyat LA, Tordoir JH, Wang Y, Wong M, Leunissen KM, van der Sande FM, Kotanko P, Kooman JP. Vascular access vulnerability in intensive hemodialysis: a significant Achilles' heel? Blood Purif. 2014;37(3):222-8. doi: 10.1159/000362106. Epub 2014 Jun 5. PMID 24902990
- [Background] Daugirdas JT, Greene T, Rocco MV, Kaysen GA, Depner TA, Levin NW, Chertow GM, Ornt DB, Raimann JG, Larive B, Kliger AS; FHN Trial Group. Effect of frequent hemodialysis on residual kidney function. Kidney Int. 2013 May;83(5):949-58. doi: 10.1038/ki.2012.457. Epub 2013 Jan 23. PMID 23344474
- [Background] Wabel P, Moissl U, Chamney P, Jirka T, Machek P, Ponce P, Taborsky P, Tetta C, Velasco N, Vlasak J, Zaluska W, Wizemann V. Towards improved cardiovascular management: the necessity of combining blood pressure and fluid overload. Nephrol Dial Transplant. 2008 Sep;23(9):2965-71. doi: 10.1093/ndt/gfn228. Epub 2008 May 5. PMID 18458032
- [Background] Wieskotten S, Heinke S, Wabel P, Moissl U, Becker J, Pirlich M, Keymling M, Isermann R. Bioimpedance-based identification of malnutrition using fuzzy logic. Physiol Meas. 2008 May;29(5):639-54. doi: 10.1088/0967-3334/29/5/009. Epub 2008 May 7. PMID 18460765
- [Background] Wizemann V, Wabel P, Chamney P, Zaluska W, Moissl U, Rode C, Malecka-Masalska T, Marcelli D. The mortality risk of overhydration in haemodialysis patients. Nephrol Dial Transplant. 2009 May;24(5):1574-9. doi: 10.1093/ndt/gfn707. Epub 2009 Jan 7. PMID 19131355
- [Background] Zoccali C, Moissl U, Chazot C, Mallamaci F, Tripepi G, Arkossy O, Wabel P, Stuard S. Chronic Fluid Overload and Mortality in ESRD. J Am Soc Nephrol. 2017 Aug;28(8):2491-2497. doi: 10.1681/ASN.2016121341. Epub 2017 May 4. PMID 28473637
- [Background] Hecking M, Moissl U, Genser B, Rayner H, Dasgupta I, Stuard S, Stopper A, Chazot C, Maddux FW, Canaud B, Port FK, Zoccali C, Wabel P. Greater fluid overload and lower interdialytic weight gain are independently associated with mortality in a large international hemodialysis population. Nephrol Dial Transplant. 2018 Oct 1;33(10):1832-1842. doi: 10.1093/ndt/gfy083. PMID 29688512
- [Background] Jotterand Drepper V, Kihm LP, Kalble F, Diekmann C, Seckinger J, Sommerer C, Zeier M, Schwenger V. Overhydration Is a Strong Predictor of Mortality in Peritoneal Dialysis Patients - Independently of Cardiac Failure. PLoS One. 2016 Jul 14;11(7):e0158741. doi: 10.1371/journal.pone.0158741. eCollection 2016. PMID 27415758
- [Background] Takahashi S. Future home hemodialysis - advantages of the NxStage System One. Contrib Nephrol. 2012;177:117-126. doi: 10.1159/000336944. Epub 2012 May 8. PMID 22613922
- [Background] Benabed A, Henri P, Lobbedez T, Goffin E, Baluta S, Benziane A, Rachi A, van der Pijl JW, Bechade C, Ficheux M. [Low flux dialysate daily home hemodialysis: A result for the 62 first French and Belgian patients]. Nephrol Ther. 2017 Feb;13(1):18-25. doi: 10.1016/j.nephro.2016.06.007. Epub 2016 Nov 18. French. PMID 27876356
- [Background] Daugirdas JT. Second generation logarithmic estimates of single-pool variable volume Kt/V: an analysis of error. J Am Soc Nephrol. 1993 Nov;4(5):1205-13. doi: 10.1681/ASN.V451205. PMID 8305648
- [Background] Wabel P, Chamney P, Moissl U, Jirka T. Importance of whole-body bioimpedance spectroscopy for the management of fluid balance. Blood Purif. 2009;27(1):75-80. doi: 10.1159/000167013. Epub 2009 Jan 23. PMID 19169022
- [Background] Leypoldt JK, Kamerath CD, Gilson JF, Friederichs G. Dialyzer clearances and mass transfer-area coefficients for small solutes at low dialysate flow rates. ASAIO J. 2006 Jul-Aug;52(4):404-9. doi: 10.1097/01.mat.0000227687.88929.08. PMID 16883120
- [Background] National Kidney Foundation. KDOQI Clinical Practice Guideline for Hemodialysis Adequacy: 2015 update. Am J Kidney Dis. 2015 Nov;66(5):884-930. doi: 10.1053/j.ajkd.2015.07.015. PMID 26498416
- [Background] Wabel P, Chamney P, Moissl U (2007) Reproducibility of bioimpedance spectroscopy for the assessment of body composition and dry weight. J Am Soc Nephrol 18: A255
- [Background] Cole, K. S., & Cole, R. H. (1941). Dispersion and absorption in dielectrics I. Alternating current characteristics. The Journal of chemical physics, 9(4), 341-351.
- [Background] Moissl UM, Wabel P, Chamney PW, Bosaeus I, Levin NW, Bosy-Westphal A, Korth O, Muller MJ, Ellegard L, Malmros V, Kaitwatcharachai C, Kuhlmann MK, Zhu F, Fuller NJ. Body fluid volume determination via body composition spectroscopy in health and disease. Physiol Meas. 2006 Sep;27(9):921-33. doi: 10.1088/0967-3334/27/9/012. Epub 2006 Jul 25. PMID 16868355
- [Background] Chamney PW, Wabel P, Moissl UM, Muller MJ, Bosy-Westphal A, Korth O, Fuller NJ. A whole-body model to distinguish excess fluid from the hydration of major body tissues. Am J Clin Nutr. 2007 Jan;85(1):80-9. doi: 10.1093/ajcn/85.1.80. PMID 17209181
- See also: épidémiologie MRC — https://www.agence-biomedecine.fr/IMG/pdf/rapport_rein_2015.pdf